CLINICAL TRIAL: NCT01333956
Title: Effects of Pregabalin on Pain After Total Knee Arthroplasty: A Randomized, Controlled, Double-Blind Trial
Brief Title: Effects of Pregabalin on Pain After Total Knee Arthroplasty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11043
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Primary Total Knee Arthroplasty
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Control (Placebo Comparator): Patients will receive 0mg of pregabalin
  Interventions: Drug: Placebo
- 50mg Arm (Experimental): Patients will receive 50mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of post-operative day (POD)14 and one capsule at bedtime POD15, POD16.
  Interventions: Drug: Pregabalin 50mg
- 100mg Arm (Experimental): Patients will receive 100mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Interventions: Drug: Pregabalin 100mg
- 150mg Arm (Experimental): Patients will receive 150mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Interventions: Drug: Pregabalin 150mg

INTERVENTIONS:
Drug: Pregabalin 50mg — Patients will receive 50mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Other Names: Lyrica
  Arms: 50mg Arm
Drug: Pregabalin 100mg — Patients will receive 100mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Other Names: Lyrica
  Arms: 100mg Arm
Drug: Pregabalin 150mg — Patients will receive 150mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Other Names: Lyrica
  Arms: 150mg Arm
Drug: Placebo — Patients will receive placebo drug with no active ingredients per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Arms: Control

SUMMARY:
Total knee arthroplasty can cause severe postoperative pain, and patients typically receive oral opioid analgesics for over 2 weeks. Side effects of pain management may impair participation in physical therapy and diminish patient satisfaction. Anecdotally, it seems that pregabalin is very helpful to patients after total knee arthroplasty. However, pregabalin can have side effects. It is not clear how much pregabalin to prescribe. Low doses may not be effective, but use of high doses may increase the incidence and severity of side effects.The purpose of this study is to determine which dosage of pregabalin is the most effective at reducing pain after knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for primary tricompartmental total knee arthroplasty with a participating surgeon
* Age 18 to 80 years old
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (primary outcome obtained via telephone call and secondary outcomes include questionnaires validated in English only)
* Patients planning on being discharged home or to a rehabilitation center that has agreed to participate

Exclusion Criteria:

* Patients younger than 18 years old and older than 80
* Patients intending to receive general anesthesia
* Allergy or intolerance to one of the study medications
* Patients with an ASA of IV
* Patients with hepatic (liver) failure
* Patients with chronic renal (kidney) failure (Defined as estimated creatinine clearance < 30 mL/min, based on recommendation that total daily pregabalin dose be reduced to 150 mg with Clcr < 30 mL/min, CLcr=[(140-age (years)] x weight (kg)x0.85 (for female patients)/[72xserum creatinine (mg/dL)])
* Patients with difficult to manage diabetes mellitus, including insulin-dependence
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Patients with major prior ipsilateral open knee surgery.
* Chronic neurontin/lyrica use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, M.D., Ph.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] YaDeau JT, Lin Y, Mayman DJ, Goytizolo EA, Alexiades MM, Padgett DE, Kahn RL, Jules-Elysee KM, Ranawat AS, Bhagat DD, Fields KG, Goon AK, Curren J, Westrich GH. Pregabalin and pain after total knee arthroplasty: a double-blind, randomized, placebo-controlled, multidose trial. Br J Anaesth. 2015 Aug;115(2):285-93. doi: 10.1093/bja/aev217. PMID 26170351

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Patients will receive 0mg of pregabalin
  Placebo: Patients will receive placebo drug with no active ingredients per dose.
- 50mg Arm: Patients will receive 50mg of pregabalin per dose.
- 100mg Arm: Patients will receive 100mg of pregabalin per dose.
- 150mg Arm: Patients will receive 150mg of pregabalin per dose.
Period: Overall Study
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Started | 30 | 30 | 30 | 30
Completed | 28 | 26 | 29 | 28
Not Completed | 2 | 4 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1
Not completed — Unable to complete study procedure | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 50mg Arm: Patients will receive 50mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
  Pregabalin 50mg: Patients will receive 50mg of pregabalin per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of POD14 and one capsule at bedtime POD15, POD16.
- Total: Total of all reporting groups
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.8) | 66.8 (6.3) | 65.1 (7.1) | 67.7 (8.1) | 66.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 13 | 23 | 68
  Male | 16 | 12 | 17 | 7 | 52
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 30 | 120
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m ^ 2] | 32 (5) | 32 (6) | 32 (6) | 30 (7) | 31.5 (2.45)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Pain assessment scale (Numeric Rating Scale) (0=no pain; 10=worst pain imaginable).
Time Frame: 2 weeks postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Patients will receive 0mg of pregabalin
  Placebo: Patients will receive placebo drug with no active ingredients per dose. 2 capsules will be taken pre-operatively. One capsule twice a day until end of post-operative day (POD)14 and one capsule at bedtime POD15, POD16.
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 28 | 26 | 29 | 28
units on a scale
  POD14 Pain score with flexion | 4 (2.3) | 4.8 (2.1) | 4.5 (2.4) | 4.0 (2.1)
  POD14 Pain score with ambulation | 3.6 (2.0) | 3.8 (1.6) | 3.5 (1.8) | 3.1 (1.9)
  POD14 Pain score at rest | 2.9 (2.3) | 2.9 (2.0) | 2.8 (1.8) | 2.7 (2.1)

2. Secondary Outcome: Opioid-Related Symptom Distress Score
Description: Opioid-Related Symptom Distress score (ORSDS) measured at POD1 and POD14. The ORSDS is a 4-point scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 12 symptoms. The symptom-specific ORSDS is the average of the 3 symptom distress dimensions. The composite ORSDS is the average of 12 symptom-specific scores. (0=low; 4=high).
Time Frame: 2 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 28 | 26 | 29 | 28
units on a scale
  ORSDS POD1 | .4 [.2 to .7] | .4 [.2 to .6] | .5 [.2 to .7] | .4 [.2 to .8]
  ORSDS POD14 | .3 [.1 to .5] | .3 [.1 to .5] | .3 [.1 to .5] | .3 [0 to .4]

3. Secondary Outcome: Self-assessed Sedation and Confusion
Description: Self-assessed sedation and confusion (POD1). Confusion Assessment Method (CAM score) (pre-operative and on POD1)
Time Frame: 1 day postoperatively
Measure: Number; unit: percentage of patients
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 29 | 29 | 29 | 29
percentage of patients
  Drowsiness POD1 [ORSDS] | 34.5 | 37.9 | 55.2 | 58.6
  Nausea POD1 [ORSDS] | 34.5 | 41.4 | 44.8 | 31.0

4. Secondary Outcome: Numeric Rating Scale (NRS)
Description: NRS Pain (pre-operative, POD1, POD3, 2 weeks, 3 months, at orthopedic visits). Neuropathic pain incidence: Leeds assessment of neuropathic symptoms and signs (LANSS) score (3 months)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 28 | 26 | 29 | 28
units on a scale
  Preop NRS Pain Score with Flexion | 4.9 [3.7 to 6] | 5.4 [4.3 to 6.5] | 3.9 [2.8 to 5.1] | 5.7 [4.4 to 7]
  POD1 NRS Pain Score with Flexion | 2.8 [1.8 to 4] | 2.9 [2 to 4] | 2.7 [1.8 to 3.3] | 2.5 [1.2 to 3.3]
  POD3 NRS Pain Score with Flexion | 3.9 [2.8 to 4.8] | 4.2 [3.5 to 5.2] | 3.6 [2.8 to 4.7] | 4.3 [3.3 to 5.3]
  POD14 NRS Pain Score with Flexion | 4 [3.4 to 5] | 4.9 [4.2 to 5.6] | 4.5 [3.7 to 5.4] | 4.2 [3.2 to 5]
  3 months NRS Pain Score with Flexion | 2 [1 to 3] | 1.9 [.9 to 2.7] | 1.7 [.7 to 1.8] | 1.8 [.9 to 2.3]

5. Secondary Outcome: Neuropathic Pain
Description: Neuropathic pain incidence: Leeds assessment of neuropathic symptoms and signs (LANSS) score (3 months). Scale of 0 to 24. Higher values represent worse outcomes.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 28 | 26 | 29 | 28
units on a scale | 0 [0 to 3] | 0 [0 to 6] | 0 [0 to 0] | 0 [0 to 3]

6. Secondary Outcome: Opioid Usage
Description: Opioid Usage (POD1, POD 3, 2 weeks, 3 months)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 28 | 26 | 29 | 28
mg
  Preop Total Opioid Use (mg) | 19 [16 to 22] | 18 [16 to 20] | 17 [15 to 19] | 18 [16 to 20]
  POD 1 Total Opioid Use (mg) | 50 [40 to 63] | 46 [35 to 57] | 57 [41 to 73] | 45 [35 to 55]
  POD 2 Total Opioid Use (mg) | 70 [57 to 85] | 60 [50 to 70] | 63 [47 to 79] | 55 [43 to 65]
  POD 3 Total Opioid Use (mg) | 55 [43 to 67] | 60 [50 to 70] | 40 [30 to 50] | 36 [30 to 42]
  POD 14 Total Opioid Use (mg) | 40 [30 to 50] | 36 [25 to 45] | 40 [30 to 50] | 45 [25 to 55]
  3 months Total Opioid Use (mg) | 0 [0 to 2] | 3 [0 to 5] | 0 [0 to 1] | 4 [0 to 6]

7. Secondary Outcome: Satisfaction
Description: Satisfaction with pain management (1-10 scale; 1 = very dissatisfied, 10 = very satisfied)
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Number analyzed (Participants) | 28 | 26 | 29 | 28
units on a scale | 9 [8 to 10] | 8 [7 to 10] | 8 [5 to 9] | 8 [6 to 9.3]

ADVERSE EVENTS:
Arm/Group | Control | 50mg Arm | 100mg Arm | 150mg Arm
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes